CLINICAL TRIAL: NCT00862745
Title: A Multi-center, Randomized, Placebo-controlled Clinical Trial Comparing Fesoterodine to Placebo in Women Diagnosed With Urge Urinary Incontinence by the 3 Incontinence Questions (3IQ). Followed by a Multi-center Open Label Clinical Cohort Study of Long-term Effects of Treatment With Fesoterodine.
Brief Title: Bringing Simple Urge Incontinence Diagnosis & Treatment to Providers (BRIDGES)
Acronym: BRIDGES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jeanette Brown, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GA0221IX
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-10

CONDITIONS: Urge Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): fesoterodine 4 mg (1 tablet) for 2 weeks with the option to increase to fesoterodine 8 mg or stay at fesoterodine 4 mg for 10 weeks for a total of 12 weeks of study medication.
  Interventions: Drug: Fesoterodine
- Control (Placebo Comparator): placebo (an identical pill that contains no medication) 1 tablet daily for 2 weeks followed by the option to increase the placebo pill daily for 10 weeks for a total of 12 weeks of study placebo medication.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Fesoterodine — Participants will be instructed to take one tablet of blinded study medication once a day, orally, for 12 weeks. They will start with a 4 mg dose of study medication and will have the option of doubling that dose after 2 or 4 weeks if they wish. At the end of the 12 week blinded trial, participants will be offered open-label fesoterodine (Toviaz™), for 9 months beginning at 4 mg with participant directed dose adjustment.
  Arms: Active
Drug: Matching Placebo — Participants will be instructed to take one tablet of blinded study medication once a day, orally, for 12 weeks. They will start with a 4 mg dose of study medication and will have the option of doubling that dose after 2 or 4 weeks if they wish. At the end of the 12 week blinded trial, participants will be offered open-label fesoterodine (Toviaz™), for 9 months beginning at 4 mg with participant directed dose adjustment.
  Arms: Control

SUMMARY:
Six hundred and thirty-six women diagnosed with urge urinary incontinence (UUI) by a three-item self-administered questionnaire (3IQ) will be randomized to 12 weeks of fesoterodine or matching placebo. The study will take place at up to 14 clinical sites in the US. All participants who complete the 12-week randomized trial will be offered open-label fesoterodine for an additional 9 months.

The hypothesis of the randomized controlled trial is that among women diagnosed with urge incontinence using the 3IQ, fesoterodine is more effective than placebo in reducing the mean number of urge incontinence episodes per day.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory females ≥ 18 years old
* Urge Urinary Incontinence (subject-reported) for ≥ 3 months prior to Screening (Visit 1)
* On the 3IQ: Response b to Question 3: During the last 3 months, did you leak urine most often: b. When you had the urge or the feeling that you needed to empty your bladder, but could not get to the toilet fast enough?
* On a 3-day bladder diary, documentation of an average of 1 UUI episode per 24 hours (3 UUI episodes in 3 days)
* Capability of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risk and benefits
* Ability to perform all procedures and tests required by the protocol
* Willingness to remain on stable medication regime for duration of the randomized controlled trial. Participants will be asked to not add new medications during the randomized controlled trial, such as diuretics and other medications which may affect their voiding pattern.

Exclusion Criteria:

* Any condition that would contraindicate their usage of fesoterodine including: hypersensitivity to the active drug (fesoterodine fumarate) and its ingredients or any of the excipients, history of urinary retention, gastric retention, uncontrolled narrow angle glaucoma, myasthenia gravis, severe hepatic impairment (Child Pugh C), severe ulcerative colitis, toxic megacolon, fistula or a hole in your bladder or rectum, birth defect leading to urine leakage, and urine leakage starting in childhood.
* Clinically significant hepatic or renal disease.
* Neurologic conditions such as stroke, multiple sclerosis, spinal cord injury, or Parkinson's disease.
* Symptomatic pelvic organ prolapse defined as participant report of feeling or seeing a bulge outside the vagina within the past 3 months.
* History of lower urinary tract/pelvic surgery (e.g. surgery for incontinence in the past 5 years, surgery in the past 6 months for prolapse or hysterectomy), intra-vesical therapy (botox), and/or bulk injections within the past 6 months.
* A known history of interstitial cystitis or a significant pain component associated with OAB symptoms, uninvestigated hematuria, urogenital cancer, interstitial or external radiation to the pelvis or external genitalia.
* Urinary tract infection (UTI) as shown by the results of the urinalysis at screening or recurrent urinary tract infection (RUTIs) defined as treatment for UTI >3 times in the last year.
* Use of any electrostimulation, bladder training, or pelvic floor exercises (with certified incontinence practitioners) within 4 weeks of Screening.
* Received study medication in any previous fesoterodine clinical trial.
* Prior failure for either efficacy or tolerability of ≥ 2 OAB medications in the last year. (failure: inadequate symptom control after two medications for a minimum of one month each)
* Has been treated within 2 weeks prior to Screening and/or is currently being treated with: - Any drug treatment for overactive bladder, including antimuscarinic OAB medications.
* Any drugs with significant anticholinergic and antispasmodic effects (see exception for tricyclic antidepressants below)
* Has started treatment with tricyclic antidepressants or estrogens within 4 weeks prior to Screening and/or is not on a stable dose.
* Intermittent or unstable use of diuretics. Treatment with diuretics initiated within 2 weeks prior to baseline is not permitted.
* Treatment with potent CYP3A4 inhibitors, such as clarithromycin, ketoconazole, and itraconazole within 2 weeks prior to Screening.
* Administration of medications capable of inducing hepatic enzyme metabolism or transport (e.g., barbiturates, rifampicin, carbamazepine, phenytoin, primidone, or St. John's Wort) in the past 30 days.
* Previously received any investigational drug within 30 days prior to trial entry.
* Alcohol and/or any other drug abuse in the opinion of the investigator.
* Participants who are pregnant, nursing, or with a positive urine pregnancy test or who are intending to become pregnant within 3 months after the completion of the trial.
* Participants that have been pregnant (> 20 weeks gestation) in the previous 6 months.
* Participants of childbearing potential who are heterosexually active but unwilling or unable to use an adequate form of contraception to prevent pregnancy during the study. Reliable contraceptive methods may include intrauterine devices (IUD), contraceptive pills of combination type, hormonal implants, injectable contraceptives or latex condoms with a spermicide.
* Participants who have any medical (including known history of major hematological, renal, cardiovascular, or hepatic abnormalities) or psychological condition or social circumstances that would impair their ability to participate reliably in the trial, or those who may increase the risk to themselves or others by participating.
* Participants who, in the opinion of the investigator, are not likely to complete the trial for whatever reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette S. Brown, MD, Principal Investigator — University of California, San Francisco
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Women & Infants' Hospital, Division of Urogynecology, Providence, Rhode Island
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Virginia-Women's Midlife Health Center, Charlottesville, Virginia

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Warsi QA, Huang AJ, Hess R, Arya LA, Richter HE, Bradley CS, Rogers RG, Myers DL, Johnson KC, Winkelman WD, Gregory WT, Kraus SR, Schembri M, Brown JS, Stone KL, Subak LL. Association of Pharmacologic Treatment of Urgency Urinary Incontinence With Sleep Quality and Daytime Sleepiness. Obstet Gynecol. 2018 Feb;131(2):204-211. doi: 10.1097/AOG.0000000000002443. PMID 29324595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general community surrounding 13 clinical sites across the United States between January 2009 and December 2009.
Pre-assignment Details: Participants screened over 4 week period.
Groups:
- Fesoterodine: fesoterodine 4 mg (1 tablet) for 2 weeks with the option to increase to fesoterodine 8 mg or stay at fesoterodine 4 mg for 10 weeks for a total of 12 weeks of study medication.
- Placebo: placebo (an identical pill that contains no medication) 1 tablet daily for 2 weeks followed by the option to increase the placebo pill daily for 10 weeks for a total of 12 weeks of study placebo medication.
Period: Randomized Control Trial
Arm/Group | Fesoterodine | Placebo
Started | 322 | 323
Completed | 284 | 284
Not Completed | 38 | 39
Period: Open-label Follow-up
Arm/Group | Fesoterodine | Placebo
Started | 268 (19 participants elected not to enter the open-label portion of the study after completing the RCT.) | 274 (10 participants elected not to enter the open-label portion of the study after completing the RCT.)
Completed | 229 | 225
Not Completed | 39 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fesoterodine | Placebo | Total
Number analyzed (Participants) | 322 | 323 | 645
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 230 | 234 | 464
  >=65 years | 92 | 89 | 181
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (14.7) | 55.9 (14.2) | 56.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 322 | 323 | 645
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 322 | 323 | 645

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Urge Urinary Incontinence Episodes at Week 12.
Time Frame: Baseline and Week 12
Population: The population analyzed included all participants receiving at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 303 | 301
episodes | -2.5 (2.5) | -1.8 (2.7)
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Null hypothesis: fesoterodine treatment is not associated with greater reduction in urgency incontinence frequency compared to placebo in women diagnosed using the 3IQ; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiple comparisons, threshold for significance is P < .05; Mean difference=Drug A minus Drug B

ADVERSE EVENTS:
Time Frame: Baseline through Week 12 (Randomized Control Trial portion of the study).
Arm/Group | Fesoterodine | Placebo
Serious Adverse Events (participants affected / at risk) | 4/322 | 4/323
Other Adverse Events (participants affected / at risk) | 148/322 | 88/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fesoterodine (N=322) | Placebo (N=323)
Hospitalized for Diabetes (Endocrine disorders) | 0 (0) | 1 (1)
Hospitalized for Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emergency Room Visit for Angina (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization for Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hosptialized for Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalization for Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fesoterodine (N=322) | Placebo (N=323)
Dry eyes/mouth/throat (Respiratory, thoracic and mediastinal disorders) | 107 (137) | 38 (54)
Constipation (Gastrointestinal disorders) | 24 (27) | 17 (17)
Headache (Nervous system disorders) | 19 (22) | 10 (10)
Cold/flu (Infections and infestations) | 21 (21) | 15 (16)
Urinary tract infection (Renal and urinary disorders) | 17 (19) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (11) | 8 (8)
Runny/stuffy nose, sinus congestion (Infections and infestations) | 8 (9) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No